CLINICAL TRIAL: NCT01337180
Title: Exposure to Aerosols and Airway Inflammation Among Workers in the Silicon Carbide Processing Industry
Brief Title: Airway Inflammation Among Workers in the Silicon Carbide Processing Industry
Status: Withdrawn | Type: Observational
Why Stopped: The industry plant from which we should recruit was closed down.
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Oslo University Hospital (Other); National Institute of Occupational Health, Norway (Other Government); University of North Carolina (Other)
Responsible Party: Principal Investigator, Anne Kristin M. Fell, Consultant, Sykehuset Telemark
Other Study IDs: 5690.14
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2013-06

CONDITIONS: Obstructive Lung Disease; Inflammation
Keywords: lung function; respiratory symptoms; dust; inflammation; prospective
MeSH Terms: conditions — Lung Diseases, Obstructive; Inflammation; Signs and Symptoms, Respiratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Induced sputum, serum, citrate- plasma, EDTA-plasma, whole blood and a PaxGene sample for DNA isolation. Cell isolation, RNA isolation and gene expression analysis. Fluid phase analyses.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Main study group: Inclusion criteria: Employment at one of the plants (SiC I) and (SiC II) in Porsgrunn. Both administrative/office workers and workers in the production and maintenance departments will be invited to participate. Non-smokers and smokers and male and female workers will be included in the main study group (study A).
  Sputum part of study: nonsmokers.

SUMMARY:
Exposure to noxious gases and particles is associated with an increased prevalence of respiratory and cardiovascular diseases. Thus, investigation of possible airway inflammation and/or systemic inflammation in workers exposed to high levels of dust is important. Silicon Carbide (SiC) Processing Inc. provides cutting fluid (slurry) for the production of solar cells and is at present the largest provider of slurry to the solar industry worldwide. In the production process, the recyclable materials (SiC), polyethylene glycol (PEG)) of the used slurry are recovered. The airborne exposure consists mainly of SiC (dust particles) and evaporation from the recycling of PEG. High levels of dust have been measured and, seventeen per cent of the measurements in the processing hall were equal to or higher than the Norwegian occupational exposure limit. Thus, assessment of possible systemic and airway effects of this exposure is of interest. A prospective design will be applied and the effects studied by means of registration of respiratory symptoms, spirometry, nitric oxide (NO) in exhaled air, induced sputum and blood sampling over a 3 year period. Exposed subjects will also be compare with non- or low exposed subjects (administrative/office workers). Efforts will be made to include all eligible subjects and to avoid drop-outs. If early signs of airway or systemic inflammation in workers or in cells are demonstrated in the study, it will be necessary to implement measures to reduce the exposure levels.

The primary aim of the present study of workers exposed to Silicon Carbide dust in the workplace is to determine whether this exposure is associated with inflammatory changes in the lungs.

The secondary aims are: - to examine possible changes in systemic inflammatory markers and - to examine changes in lung function among Silicon Carbide processing workers during a period of 3 years. Possible changes in lung function will be monitored by spirometry and gas diffusion measurements (study A). Airway inflammatory responses and changes in circulating inflammatory markers will be assessed by examination of the induced sputum samples and blood samples every 6th month in a subgroup of workers (study B).

DETAILED DESCRIPTION:
Does exposure to aerosols induce airway inflammation and/or a systemic inflammatory response in workers in the silicon carbide (SiC) processing industry?

As yet, no human studies describing the health effects from exposure during recycling of slurry containing SiC and/or PEG have been reported. However, there are several studies that may be relevant which assess the health effects of other particles. It has been demonstrated that small particles penetrate further into the lungs than larger particles and thereby have stronger irritating properties [2]. Results from 2 experimental studies where the effect variables were lung function, organ weights and characteristics of broncho-alveolar lavage (BAL) [3, 4] indicate that SiC dust and PEG itself are probably relatively inert. However, in a third study it was demonstrated that SiC particles have the potential to stimulate test cells (murine macrophage cell line and human osteoblast-like cell line) to produce inflammatory signal substances (tumour necrosis factor (TNF)-alfa), indicating possible inflammatory responses in the lungs [5]. Furthermore, it is thought that the total amount of inhaled dust is important ("overload") even if the substance itself is relatively inert [6]. Repeated high exposures (peaks) may act as a reinforcing factor.

Because there are few previous studies, and the available data are conflicting, there is a need for more knowledge about the association between health effects and exposure to particles in general and to exposure in the SiC processing industry in particular.

Our hypothesis is that airway inflammation may be induced by exposure to SiC particles and would probably be detectable as increased levels of inflammatory cells and soluble inflammatory markers in the sputum and blood samples from non-smoking, asymptomatic workers.

The primary aim of the present study of workers exposed to SiC dust in the work-place is to determine whether this exposure is associated with inflammatory changes in the lungs.

The secondary aims are:

* to examine possible changes in systemic inflammatory markers, and
* to examine changes in lung function among SiC-processing workers over a period of 3 years.

Possible changes in lung function will be monitored by spirometry measurements (study A). Airway inflammatory responses and changes in circulating inflammatory markers will be assessed by examination of the induced sputum samples and blood samples in a subgroup of workers (study B).

General value An important goal of the study is to provide knowledge that can be important for workers who are exposed to particles and aerosols in the SiC-processing industry or other industries processing SiC and/or PEG. The study may also be relevant to workers in other industries with dusty environments given the possible "overload" mechanisms. The study could possibly also have the potential to provide additional knowledge about effects of exposure to similar particles e.g from air pollution. Because few former studies have used induced sputum in a prospective design, such studies are of particular interest.

If early signs of lung inflammation or a decrease in lung function are demonstrated in the present study, it will be necessary to implement additional measures to reduce the dust levels in this industry; e.g., through enclosure of processes. The investigators believe that the results from this study together with the existing knowledge of inflammatory effects associated with occupational exposure to particles may be relevant for the prevention of chronic respiratory disease.

III - Study design and methods Study population In the present study, the effects of exposure to aerosols on airway inflammation and systemic inflammation will be investigated by means of spirometry, FeNO, induced sputum and blood sampling over a three-year period.

Study A: The whole group of workers will complete a questionnaire on respiratory symptoms and undergo spirometry at baseline, and again after 3 years. All former workers will be contacted and asked to complete a questionnaire to assess the proportion of workers resigning because of (or partly because of) health effects. These workers will also be invited to undergo an examination of lung function (spirometry). This is to ensure that all workers ever employed are included in the study population.

Study B: A subgroup comprising non-smokers will in addition be followed with blood samples, induced sputum tests and exposure measurements every 6 months over the same time period.

Controls: Exposed subjects will be compared with non- or low-exposed subjects (administrative/office workers). In addition to the prospective study, the investigators will compare the baseline findings from the sputum and blood samples with those from already established external control groups from previous studies on healthy non-exposed workers and from cement production workers from the same geographic area [7].

Exposure-response analyses: Workers will be divided into groups with different exposure levels in order to study exposure-response trends of the measured agents in the exposed population (this design is less vulnerable to selection effects).

Baseline examinations will be repeated for all subjects and for the sputum subgroup. Detailed, validated questionnaires will record the medical history, relevant illnesses, use of medications, occupational history as well as present exposures.

Spirometry will allow registration of lung function and FeNO measurements the monitoring of possible airway inflammation.

A group-based strategy will be applied for the collection of exposure measurements at baseline and at follow-up (3 years) for the subjects not included in the sputum part of the study.

Induced sputum collection will be applied to detect possible changes in inflammatory cells and soluble markers from the airways.

Blood analysis will be collected to examine possible changes in circulating inflammatory markers and their association to exposure.

All participants in the sputum subgroup will carry individual exposure measurement.

The employees who leave the cohort will contribute with data while they are employed (defined as time-at-risk) and a drop-out test will be performed to determine whether they experienced work-related respiratory symptoms or diseases. New employees will be included during the study period and assigned a time-at-risk equal to their time of exposure.

Exposure measurement and assessment The dust/aerosol samples will be collected with the use of thoracic and inhaled respirable cyclones to estimate the doses for the deposition in the bronchi and in the alveoli.

Validity Factors that may affect lung function and inflammatory markers in sputum Age, height, BMI and sex will be recorded for the study. Height in meters will be entered into the computer program for calculating spirometry values. Weight (body mass index) affects lung function and will be measured before the examination. The investigators will also record possible acute respiratory infections during the preceding 12 months. An upper respiratory infection during the preceding three weeks may affect the level of inflammatory cells and markers in sputum.

There is a possibility that very early inflammatory effects among these workers could be succeeded by adaptation and thereby reduction of effects. In this case, the inflammatory response at some time after employment could be smaller than observed initially. This may lead to underestimation of effects. The investigators consider that a dynamic cohort design including only subjects exposed for the first time in this industry is not feasible. However, a follow-up of three years is considered sufficient to detect clinically relevant changes. The cohort in this study will also have a relatively short prior employment in the industry because the plants were opened in 2006 and 2009. Spirometry screening of all workers, performed during the first days of employment at the local health services, is available. These will be compared with the baseline recordings to evaluate possible effects prior to inclusion in the present study.

Statistical analysis and study power

The associations to be studied are individual changes in the effect variables:

* the trend over the study period (study A: baseline and 36 months for the whole group of workers; study B for the sputum subgroup: baseline, 6, 12, 24 and 36 months), and
* between exposed and controls (exposed and unexposed/administrative staff/office workers) at baseline and differences in trend during the study period.

T tests will be used to compare cases and controls at baseline for normally distributed variables, and a Mann-Whitney test for non-normally distributed variables. Where multiple tests are to be conducted, ANOVA and Kruskal-Wallis tests will be applied prior to the pairwise comparisons to determine the overall significance level.

Multiple regression models with adjustment for age, sex, smoking habits and other relevant factors for each analysis will be applied when adjusting for other factors at baseline.

To analyse the repeated measures, general linear models (GLM) and mixed models will be used.

The power calculations are based on clinically interesting differences in percentage of neutrophils and spirometry values. The study is designed to include at least 20 participants in each group based on a power estimate of 90%, which assumes a 95% significance level, to detect a true difference in the percentage neutrophils between two tests of at least 16%. Power calculation for FEV1 and FVC% of predicted: if the goal is to detect a difference of 1.5% in FEV1 and FVC% predicted, then given a standard deviation of 5% the sample must consist of 117 persons in each group. This will ensure 90% power to detect a difference at the 5% significance level.

It is expected that the response rate among non-smokers will allow approximately 40 employees and 20 unexposed workers to be included in the sputum part of the study (study B). Based on the power calculations, prior experience and published studies, this will be enough to detect a difference in development between the two groups of the expected magnitude. In total, 150 workers are employed at SiC I and II (to be included in study A). It is planned to include the employees at Glomfjord (Nordland) SiC processing if the sample size from Porsgrunn is not sufficient. To ensure sufficient unexposed workers, the neighbouring Renewable Energy Corporation (REC) plant will be used to recruit controls if needed. The REC plant started production at about the same time and has a similar work-force to the study group.

VI - Ethical aspects It is considered that the purpose of the study and the methods being used do not violate generally accepted ethical values. Participation in the project is voluntary. Collection of biological material and information will take place with the participants' consent. All participants will sign consent forms after receiving written information about the survey. Participants will at any time have the opportunity to withdraw from the study without giving a reason.

According to an agreement with the SIC- processing, the research fellow and project group can freely publish the results of the survey. The project is not financially dependent on grants from the industry, and the industry (SIC) financing of the project is limited to the exposure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Employment at SiC plant in Porsgrunn;

Exclusion Criteria for sputum study:

* smoking
* active airway infection or less then 3 weeks after recovery
* active allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employment at one of the plants (SiC I) and (SiC II) in Porsgrunn. Both administrative/office workers in the production and maintenance departments will be invited to participate. Non- smokers and smokers and male and female workers will be included in the main study group. Only non- smokers will be included in the sputum part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Johny Kongerud, professor, Study Director — Oslo University; Oslo University Hospital; Berit Bakke, PhD, Principal Investigator — National Institute of Occupational Health; Anne Kristin M Fell, MD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Sykehuset Telemark, Skien, Telemark, Norway

REFERENCES:
- [Background] Sioutas C, Delfino RJ, Singh M. Exposure assessment for atmospheric ultrafine particles (UFPs) and implications in epidemiologic research. Environ Health Perspect. 2005 Aug;113(8):947-55. doi: 10.1289/ehp.7939. PMID 16079062
- [Background] Bruch J, Rehn B, Song H, Gono E, Malkusch W. Toxicological investigations on silicon carbide. 1. Inhalation studies. Br J Ind Med. 1993 Sep;50(9):797-806. doi: 10.1136/oem.50.9.797. PMID 8398873
- [Background] Bruch J, Rehn B, Song W, Gono E, Malkusch W. Toxicological investigations on silicon carbide. 2. In vitro cell tests and long term injection tests. Br J Ind Med. 1993 Sep;50(9):807-13. doi: 10.1136/oem.50.9.807. PMID 8398874
- [Background] Allen M, Butter R, Chandra L, Lettington A, Rushton N. Toxicity of particulate silicon carbide for macrophages, fibroblasts and osteoblast-like cells in vitro. Biomed Mater Eng. 1995;5(3):151-9. PMID 8555965
- [Background] Fell AK, Sikkeland LI, Svendsen MV, Kongerud J. Airway inflammation in cement production workers. Occup Environ Med. 2010 Jun;67(6):395-400. doi: 10.1136/oem.2009.047852. Epub 2009 Oct 22. PMID 19854695
- [Background] Toren K, Brisman J, Jarvholm B. Asthma and asthma-like symptoms in adults assessed by questionnaires. A literature review. Chest. 1993 Aug;104(2):600-8. doi: 10.1378/chest.104.2.600. PMID 7802735
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Macintyre N, Crapo RO, Viegi G, Johnson DC, van der Grinten CP, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, Gustafsson P, Hankinson J, Jensen R, McKay R, Miller MR, Navajas D, Pedersen OF, Pellegrino R, Wanger J. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J. 2005 Oct;26(4):720-35. doi: 10.1183/09031936.05.00034905. No abstract available. PMID 16204605
- [Background] Sikkeland LI, Haug T, Stangeland AM, Flatberg G, Sostrand P, Halvorsen B, Kongerud J. Airway inflammation in paper mill workers. J Occup Environ Med. 2007 Oct;49(10):1135-42. doi: 10.1097/JOM.0b013e31814b2e87. PMID 18000418
- [Background] Pin I, Gibson PG, Kolendowicz R, Girgis-Gabardo A, Denburg JA, Hargreave FE, Dolovich J. Use of induced sputum cell counts to investigate airway inflammation in asthma. Thorax. 1992 Jan;47(1):25-9. doi: 10.1136/thx.47.1.25. PMID 1539140
- [Background] Sikkeland LI, Kongerud J, Stangeland AM, Haug T, Alexis NE. Macrophage enrichment from induced sputum. Thorax. 2007 Jun;62(6):558-9. doi: 10.1136/thx.2006.073544. No abstract available. PMID 17536036
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806